CLINICAL TRIAL: NCT06124196
Title: Wearable Technology to Evaluate Hyperglycemia and Heart Rate Variability in Duchenne Muscular Dystrophy
Brief Title: Wearable Technology to Evaluate Hyperglycemia and HRV in DMD
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jaclyn Tamaroff, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 231636
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; heart failure; cardiomyopathy; hyperglycemia; heart rate variability; remote; controls
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Heart Failure; Cardiomyopathies; Hyperglycemia | interventions — Wearable Electronic Devices; Exercise Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case - DMD: 40 male individuals with DMD
  Interventions: Device: wearable technology
- Controls: 40 matched controls (gender, age ± 1 year, BMI category, self-reported race/ethnicity).
  Interventions: Device: wearable technology

INTERVENTIONS:
Device: wearable technology — Three wearable devices
  Other Names: Continuous glucose monitor (CGM): The Dexcom G6 Pro Continuous Glucose Monitoring System (Dexcom G6 Pro System); Holter Monitor: Body Guardian Mini Remote Monitoring System; Physical activity and sleep monitor: ActiGraph GT9X accelerometers

SUMMARY:
Duchenne muscular dystrophy (DMD) is an X-linked disorder that causes muscle wasting, cardiopulmonary failure, and premature death. Heart failure is a leading cause of death in DMD, but substantial knowledge gaps exist regarding predisposing risk factors. In the general population, hyperglycemia, insulin resistance, and decreased heart rate variability (HRV; reflecting autonomic dysfunction) are associated with cardiomyopathy (CM). It is unclear whether these factors are associated with DMD-CM. Closing this knowledge gap may lead to novel screening and therapeutic strategies to delay progression of DMD-CM, now the leading cause of death in patients with DMD. Despite risk factors for hyperglycemia, including the use of glucocorticoids (GCs), sarcopenia, obesity, and reduced ambulation, little is known regarding glucose abnormalities in DMD. Some of these same risk factors, along with the distance needed to travel for specialty care, present significant barriers to research participation and clinical care for individuals with DMD. Remote wearable technology may improve research participation in this vulnerable population. Therefore, this study will leverage remote wearable technologies to overcome these barriers and define the relationship between dysglycemia and DMD-CM.

The goal of this remote study is to evaluate rates of hyperglycemia in individuals with DMD compared to control participants using continuous glucose monitors, and to determine the relationship between hyperglycemia and heart rate variability. Participants will utilize continuous glucose monitors, cardiac monitors, and activity monitors to evaluate glucose levels, heart rate, activity, and sleep.

DETAILED DESCRIPTION:
This study is a critical first step in evaluating hyperglycemia in DMD and the relationship to autonomic dysfunction. Our findings will help establish screening guidelines and provide a basis for intervention studies targeting glycemia in DMD. Additionally, this study, along with other ongoing studies (Wearable Technology to Evaluate Hyperglycemia and Heart Rate Variability in Duchenne Muscular Dystrophy - longitudinal aim) will establish wearable technology as investigational tools, for potential use in future clinical trials, in individuals with DMD and neuromuscular diseases.

Study Population: This study will include approximately 40 participants with DMD and 40 age/gender/BMI category, race and ethnicity matched participants without DMD.

DMD is an X-linked disorder affecting approximately 1/3500-6000 males and 1/50 million females. Therefore, only males will be included in this study.

Study Enrollment Period: Expected duration of the study is 6 years.

Study procedures (remote or in-person):

* Medical history and record review
* Continuous Glucose Monitor (CGM) A CGM sensor (Dexcom Pro, Dexcom Inc, San Diego, CA) will be placed on the abdomen of each participant during the study visit or sent to the participant's home. If the CGM sensor is placed remotely, the process of CGM placement will be reviewed over a video call with study staff. Participants will wear the CGM for up to 10 days (blinded) then return it via pre-paid envelope. The CGM collects glucose data every 5 minutes. Participants will be offered an optional "skin grip" adhesive (Skin Grip, Bountiful, UT) that they have the option to place over the CGM sensor to help keep it in place.
* Activity Monitoring (ActiGraph) Activity and sleep duration will be measured over 1-week using the ActiGraph accelerometers (ActiGraph, LLC, Pensacola, FL). Participants are instructed to wear the monitors on their dominant wrist for 7 days, 24 hours per day. Data is collected via ActiGraph at a rate of 40Hz and analyzed in 15-second epochs (ActiLife version 6.4 software, Pensacola, FL). For both activity and sleep parameters, the minimum valid wear time to utilize the data is 1 weekend day/night and 3 weekday days/nights with at least 6 hours of wear time per day/night.
* Holter (cardiac) Monitoring An extended-wear Holter monitor (Body Guardian Mini, Preventice, Rochester, MN) will be placed by study personnel during in person visits or participants at home. Participants will wear the monitor for 7 days at the same time they are wearing the CGM and ActiGraph. HRV is automatically calculated by the software.
* Diary/electronic survey Participants will be asked to complete a brief diary/survey response (approximately 5-minute survey twice daily). The REDCap survey diary will be texted to participants in the morning and evening via REDCap/Twilio. The diary will include questions related to sleep, activity, and food intake. Participants will be asked to complete the survey for the 7 days that they are wearing both the ActiGraph and the CGM.

ELIGIBILITY:
CASE, DMD inclusion criteria:

* Male
* Age ≥10years
* Clinical phenotype of DMD confirmed with muscle biopsy or genotype.
* Informed consent for individuals ≥18 years
* Parent/guardian informed consent and child assent for individuals < 18 years

CASE, DMD exclusion criteria:

* Refusal to participate.
* Diagnosis of diabetes prior to the study and/or taking insulin or other anti-diabetic drug therapy in < 4 weeks prior to treatment
* Use of a pacemaker, Implantable cardioverter-defibrillator (ICD), or other implanted device
* Unable to comply with study procedures, in the opinion of the investigator.

CONTROL inclusion criteria:

* Male
* Age ≥10years
* Informed consent for individuals ≥18 years
* Parent/guardian informed consent and child assent for individuals < 18 years
* BMI matched by Centers for Disease Control and Prevention (CDC) category (underweight, normal, overweight, obese) to cases.
* Self-reported race/ethnicity matched to cases.
* No known evidence of diabetes, impaired fasting glucose, or impaired glucose tolerance:
* For individuals (all ≥10 years) of age with obesity, we anticipate that they will have hemoglobin A1c (HbA1c) screening based on American Academy of Pediatrics (AAP) recommendations.
* Participants will be included if they have a normal HbA1c (< 5.7%) or if they have an elevated HbA1c (5.7-6.4%) with no evidence of impaired fasting glucose or impaired glucose tolerance on clinically obtained oral glucose tolerance tests (OGTT) (e.g., fasting glucose <100mg/dL and 2-hour glucose <140mg/dL).

CONTROL, exclusion criteria:

* Refusal to participate.
* Diagnosis of diabetes prior to the study and/or taking insulin or other anti-diabetic drug therapy in < 4 weeks prior to treatment
* Use of a pacemaker, Implantable cardioverter-defibrillator (ICD), or other implanted device
* Unable to comply with study procedures, in the opinion of the investigator.
* Diagnosis of DMD or Becker muscular dystrophy

Min Age: 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — DMD is an X-linked disorder affecting approximately 1/3500-6000 males and 1/50 million females. Therefore, only males will be included in this study.
  Investigators will not obtain confirmation of biological sex and accept all participants as they self-identify.
Study Population: Case: 40 adolescent and young adult males with DMD Control: 40 adolescent and young adult males without DMD
  DMD affects about 1/3500-6000 males and 1/50million females, therefore only male participants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Rate of hyperglycemia | once over 10 days
  number of glucose measurements ≥140mg/dL over total number of glucoses compared between individuals with and without DMD
Standard deviation of the mean R-to-R segment (SDANN) | once over 7 days
  correlation of rate of hyperglycemia and SDANN, which reflects heart rate variability

SECONDARY OUTCOMES:
Coefficient of variation on CGM | once over 10 days
  variability of glucose levels on CGM measured by COV compared between individuals with and without DMD
Rate of significant hyperglycemia | once over 10 days
  number of glucose measurements ≥200mg/dL over total number of glucoses compared between individuals with and without DMD
Activity level - measured by ActiGraph | once over 7 days
  Time spent in sedentary, low intensity, and moderate to vigorous physical activity. Physical activity will be measured over 1-week using the ActiGraph GT9X accelerometers (ActiGraph, LLC, Pensacola, FL).
Standard deviation of normal R to R intervals (SDNN) | once over 7 days
  correlation of rate of hyperglycemia and SDNN

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Tamaroff, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No